CLINICAL TRIAL: NCT06485362
Title: Use of Thermography for the Prevention and Diagnosis of Diabetic Foot
Status: Not yet recruiting | Type: Observational
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, ANA MARIA RAYO PEREZ, Principal Investigator, University of Seville
Other Study IDs: TERMOGRAPGY-DIABETICFOOT
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Foot; Diabetic Neuropathies; Diabetic Angiopathy
Keywords: diabetic foot; neuropaty; angiopaty; termography
MeSH Terms: conditions — Diabetic Foot; Diabetic Neuropathies; Diabetic Angiopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Healthy subjects will have thermographic images of both feet taken in multiple views
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy patients: Subjects healthy will rest barefoot for 15 minutes in a room at constant temperature (22-24°C).
  Thermographic images of both feet will be taken in multiple views (dorsal, plantar, lateral).
  Images will be analyzed to identify temperature differences between different areas of the foot and between study groups.
  Interventions: Diagnostic Test: Termography
- diabetic foot patients: Subjects with diabetic foot, diagnosed with diabetes mellitus for more than 5 years, will rest barefoot for 15 minutes in a room at a constant temperature (22-24°C).
  Thermographic images of both feet will be taken in multiple views (dorsal, plantar, lateral).
  The images will be analyzed to identify temperature differences between different areas of the foot and between the study groups.
  Interventions: Diagnostic Test: Termography

INTERVENTIONS:
Diagnostic Test: Termography — Thermographic images of both feet will be taken in multiple views (dorsal, plantar, lateral).

SUMMARY:
Diabetic foot is a serious complication of diabetes mellitus that can lead to ulcerations, infections and, in extreme cases, amputations. Early detection of changes in skin temperature can help prevent these complications. Infrared thermography is a noninvasive technique that allows the visualization and quantification of skin temperature and could be an effective tool for the early detection of alterations in diabetic foot.

Objective

To evaluate the effectiveness of infrared thermography in the early detection and diagnosis of diabetic foot, comparing the temperatures of the feet of healthy subjects and subjects with diabetic foot.

DETAILED DESCRIPTION:
Significant differences in foot temperatures are expected to be found between subjects with diabetic foot and healthy subjects. It is anticipated that areas of the foot at higher risk of ulceration in subjects with diabetic foot will show higher temperatures due to inflammation and changes in blood perfusion.

The results of the study could validate the use of thermography as an early detection and monitoring tool in patients at risk of developing diabetic foot. This could allow early and personalized interventions to prevent serious complications.

ELIGIBILITY:
Inclusion Criteria:

Subjects of both sexes. Age between 40 and 80 years. Diagnosis of type 1 or type 2 diabetes mellitus (for the case group). Absence of acute inflammatory diseases in the control group. Signed informed consent.

Exclusion Criteria:

Skin diseases that affect the interpretation of thermography. Recent treatment with medications that affect peripheral circulation. History of lower limb amputation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects or those with type 2 diabetes mellitus for more than 5 years who wish to participate in the study voluntarily, who will undergo a thermography of both feet.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Temperature maximun | One measurement will be taken at the start of the study and another measurement the following year.
  Maximum foot temperatures
Temperature minimum | One measurement will be taken at the start of the study and another measurement the following year.
  Minimum foot temperatures

CONTACTS AND LOCATIONS:
Overall Officials: RAQUEL GARCIA DE LA PEÑA, DOCTOR, Principal Investigator — University of Seville
Locations (1):
- University of Seville, Seville, Spain

IPD SHARING:
Plan to Share IPD: No